CLINICAL TRIAL: NCT04091308
Title: Individualized Physical Exercise Training and Enhanced Protein Intake in Older Citizens During Municipality-based Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Absalon (Other)
Collaborators: University of Southern Denmark (Other); Sundhed og Træning, Slagelse Municipality (Unknown); Arla Foods (Industry); Danish Council for Independent Research (Other); Association of Danish Physiotherapists (Other)
Responsible Party: Principal Investigator, Sanel Teljigovic, Senior lecturer, PhD-student, University College Absalon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8045-00052B; SJ-758 (Other: Ethics Committee, Region Zealand, Denmark)
Record Dates: First submitted 2019-09-04; First posted 2019-09-16 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Rehabilitation
Keywords: Exercise; Protein supplementation; Physical exercise training
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (Active Comparator): Usual care involves physiotherapeutic rehabilitation in an unknown format, and will, therefore, be monitored closely and described accordingly.
  Interventions: Other: Usual Care
- Usual Care with Protein Supl. (Experimental): Usual care involves physiotherapeutic rehabilitation in an unknown format, and will, therefore, be monitored closely and described accordingly.
  Interventions: Other: Usual Care with Protein Supplementation
- Individualized Physical Exercise Training with Protein Supl. (Experimental): This group is also called EXER group, and will receive individually tailored physical exercise programs, based on their strength and weaknesses from the baseline testing.
  Interventions: Other: Individualized Physical Exercise Training with Protein Supplementation

INTERVENTIONS:
Other: Usual Care — Usual care involves physiotherapeutic rehabilitation in an unknown format, and will, therefore, be monitored closely and described accordingly.
  Arms: Usual Care
Other: Usual Care with Protein Supplementation — The intake of protein supplementation (ARLA PROTINO) will be consumed by participants in the form of protein-enriched yogurts for easy consumption two times daily, with each bottle containing 14 g of protein.
  Other Names: ARLA PROTINO
  Arms: Usual Care with Protein Supl.
Other: Individualized Physical Exercise Training with Protein Supplementation — Besides getting prescribed individualized physical exercise training programs, this group will consume protein supplementation (ARLA PROTINO) in form of protein enriched yogurts for easy consumption, two times daily, with each bottle containing 14 g of protein.
  Other Names: ARLA PROTINO
  Arms: Individualized Physical Exercise Training with Protein Supl.

SUMMARY:
The study will investigate if: 1) individualized physical exercise training in combination with extra protein intake can increase measures on all three ICF-levels? 2) extra protein intake alone increases outcomes of usual care treatment?

DETAILED DESCRIPTION:
Successful rehabilitation of the growing number of elderly citizens can lead to preservation of functional independence and improvement in the quality of life.

The aim of the study is to investigate the effect of an individually tailored physical exercise training program combined with increased protein intake in order to improve measures on all three ICF levels (International Classification of Functioning, Disability, and Health). By conducting the study in a real-life clinical setting, research is translated into practice involving health professionals and the target group in the development of new knowledge on how to enhance the outcome of rehabilitation, thereby increasing the overall capacity of the elderly citizen, and decreasing the expenditure of health-services.

ELIGIBILITY:
Inclusion Criteria:

All citizens that are referred to the health/rehabilitation center age 65 years and older from Slagelse municipality will be invited to a screening interview with a physiotherapist after which the participant will be asked to join the study if not subject to one of the following exclusion criteria's:

Exclusion Criteria:

* inability to speak or read Danish,
* renal diseases,
* active cancer,
* upper or lower limp amputations,
* milk/lactose allergy or intolerance,
* hypertension >180/110,
* pacemaker/other implanted electrical stimulants (due to Bio-Impedance Analysis),
* progressive somatic or psychiatric diseases which can affect the course of training,
* referred to rehabilitation primarily due to gynecological and neurological conditions (apoplexies) or surgeries where movement restrictions are recommended,
* daily medication that may have an impact on muscle protein synthesis,
* alcohol intake greater than 14 units per week,
* discouragement from a general practitioner.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Short Musculoskeletal Function Assessment (SMFA) - Dysfunction Index | Change from: baseline to 3 months (primary endpoint) and 12 months
  Self reported

SECONDARY OUTCOMES:
Mean change from baseline in mobility with The New Mobility Score | Change from: baseline to 3 months and 12 months
  The New Mobility Score assesses the patient's walking function inside, outside, and during shopping. Including whether a walking aid is used. The NMS provides a composed score of the participants' mobility. Each question is scored between 0-3 points, depending on the degree of help. The total possible score is between 0 and 9 points.
Mean change from baseline in the PRISMA-7 score | Change from: baseline to 3 months and 12 months
  The PRISMA-7 questionnaire is composed of seven items and is used to indicate frailty among participants - each question scores either 0 or 1 points. The total possible score is between 0 and 7 points.
Mean change from baseline in the Tilburg Frailty Scale score | Change from: baseline to 3 months and 12 months
  The Tilburg Frailty Scale is a questionnaire with a bio-psycho-social approach, which measures frailty. It is composed of 15 multidimensional questions, regarding the physical, psychological, and social aspects of human functioning.
  Scoring range is between 0-15 points.
Mean change from baseline in health-related quality of life on SF-36 | Change from: baseline to 3 months and 12 months
  The SF-36 is a generic questionnaire that measures health-related quality of life in the past four weeks. The questionnaire consists of 36 questions which are divided into eight sub-scales and summarized in 2 sum scores.
Measure of pain, physical activity level and educational level | Change from: baseline to 3 months and 12 months
  A survey with self-formulated questions regarding name, sex, personal ID (CPR number), educational level, the region of pain the last three months (marked on a body chart), pain intensity at the site of pain, and physical activity level will also be collected.
Mean change from baseline in weight | Change from: baseline to 3 months and 12 months
  Weight (in kilograms). Weight and height will be combined to report BMI in kg/m^2.
Measure of height at baseline | Baseline
  Height (in meters). Weight and height will be combined to report BMI in kg/m^2.
Mean change from baseline in blood pressure | Change from: baseline to 3 months and 12 months
  Systolic and diastolic blood pressure (mmHg) will be measured using the Omron HBP 1100 blood pressure and resting heart rate monitor.
Mean change from baseline in resting heart rate | Change from: baseline to 3 months and 12 months
  Resting heart rate (in beats per minute) will be measured using the Omron HBP 1100 blood pressure and resting heart rate monitor.
Mean change from baseline in body composition measured with a bioimpedance device | Change from: baseline to 3 months and 12 months
  The electrical bioimpedance device used in the present study to measure changes in body composition is the "Tanita 9MC-780U Multi Frequency Segmental Body Composition Analyzer".
  Lean body mass (in kilograms), fat percentage (described as a percentage of the total body mass), total body water (described as a percentage of the total body mass), a visceral fat indicator will be reported
Mean change from baseline in the basic metabolic rate (BMR) | Change from: baseline to 3 months and 12 months
  BMR will be estimated by a bioelectrical impedance analysis device "Tanita 9MC-780U Multi Frequency Segmental Body Composition Analyze".
Mean change from baseline of Waist-To-Hip ratio | Change from: baseline to 3 months and 12 months
  The circumference of the waist (in centimeters) will be divided with the circumference of the hip (in centimeters) to report the Waist-to-hip ratio.
Mean change from baseline in maximal isometric voluntary contraction of leg extension | Change from: baseline to 3 months and 12 months
  A maximal isometric voluntary contraction (in newtons) for knee extension will be performed using a strain gauge.
Mean change from baseline in handgrip strength | Change from: baseline to 3 months and 12 months
  The handgrip strength (in kilograms) will be measured using a hydraulic handgrip dynamometer (SAEHAN).
Mean change from baseline in leg press strength | Change from: baseline to 3 months and 12 months
  Five repetitions maximum (RM) strength tests will be performed in the leg press (in kilograms) to calculate 1 RM.
Mean change from baseline in knee extension strength | Change from: baseline to 3 months and 12 months
  Five repetitions maximum (RM) strength tests will be performed in knee extension (in kilograms) to calculate 1 RM.
Mean change from baseline in calf extension strength | Change from: baseline to 3 months and 12 months
  Five repetitions maximum (RM) strength tests will be performed in the calf extension (in kilograms) to calculate 1 RM.
Mean change from baseline in function measured with the 2 minutes walk test (2MWT) | Change from: baseline to 3 months and 12 months
  The 2MWT will measure the distance (in meters) a person can walk in 2 minutes. Gaits speed will be calculated by dividing the covered distance with the time (120 seconds).
Mean change from baseline in heart rate during 2 minutes walk test (2MWT) | Change from: baseline to 3 months and 12 months
  Heart rate (in BPM) will be measured (using the Apple Watch serie 5) before and right after the 2MWT.
Mean change from baseline in heart rate before and after the 2 minutes walk test (2MWT) | Change from: baseline to 3 months and 12 months
  Heart rate (in BPM) will be measured (using the Apple Watch serie 5) before and right after the 2MWT.
Mean change from baseline in The Borg Rating of Perceived Exertion before and after the 2 minutes walk test (2MWT) | Change from: baseline to 3 months and 12 months
  The Borg Rating of Perceived Exertion will be used to estimate the activity intensity before and right after the 2MWT.
Mean change from baseline in function measured with the Timed Up and Go test (TUG) | Change from: baseline to 3 months and 12 months
  Time is noted (in seconds) on how long it takes to get up from a chair, walk 3 meters, turn around and go back to the chair and sit down again.
Mean change from baseline in balance measured with the Tandem test | Change from: baseline to 3 months and 12 months
  A measure of static balance will be performed using a Tandem test. The participants will be tested in three positions for 10 seconds each (feet together, semi tandem and full tandem). Time is noted (in seconds) for how long the participant can stand in each position.
Balance and reaction time for upper and lower extremity | Change from: baseline to 3 months and 12 months
  Measures for balance and reaction time will be collected using the "Fysiometer," and the protocols within the "Fysiometer" software will be followed.
Protein and energy intake | Change from: baseline, week 3, week 6, week 9, 3 months and 12 months
  During the 12-week intervention period, protein and energy intake will be estimated based on the average of four 24-hour dietary recall interviews, either by home visits or by phone. Dietary interviews will also be conducted at 12 month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Sanel Teljigovic, PhD student, Principal Investigator — University College Absalon & University of Southern Denmark
Locations (1):
- Sundhed og Træning, Slagelse, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data collected during the project period will be sent to "The Danish National Archives" https://www.sa.dk/en/
Supporting Information: Study Protocol
Time Frame: Data will be available immediately after it is submitted to the Danish National Archives.
Access Criteria: Data is managed by the Danish National Archives and can be disclosed according to the Danish "notes of archive act / LBK no. 1201 from 28/09/2016".
URL: https://www.sa.dk/en/

REFERENCES:
- [Derived] Teljigovic S, Sogaard K, Sandal LF, Dalager T, Nielsen NO, Sjogaard G, Holm L. Individualised physical exercise training and enhanced protein intake in older citizens during municipality-based rehabilitation: protocol for a randomised controlled trial. BMJ Open. 2020 Nov 26;10(11):e041605. doi: 10.1136/bmjopen-2020-041605. PMID 33243811